CLINICAL TRIAL: NCT04174313
Title: Ventilator-induced Lung Injury Vortex in Patients With SARS-CoV-2
Acronym: VILIVORTEX
Status: Completed | Type: Observational
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, Head of Intensive Care Unit at Hospital El Cruce, Hospital El Cruce
Other Study IDs: Nestor Pistillo
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Results first posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: ARDS; Mechanical Ventilation Complication; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VILI VORTEX and No VILI VORTEX: Measurement of pulmonary pressures and volumes in the same patient
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — Mechanical variables and PaO2/FiO2 were registered daily for 14 days or until initiating assisted ventilation. These data were obtained in passive mechanical conditions.
  Ventilator-induced lung injury vortex was defined as a progressive increase in driving pressure (ΔP) as Vt remained constant or even decreased.
  Refractory hypoxemia was defined as PaO2/FiO2 <100 despite the optimization of mechanical ventilation and prone positioning.
  Other Names: Transpulmonary pressures (TP) will be measured

SUMMARY:
The concept of Ventilator-induced Lung Injury Vortex (VILI vortex) has recently been proposed as a progressive lung injury mechanism in which the alveolar stress/strain increases as the ventilable lung "shrinks" (1). This positive feedback inexorably leads to the acceleration of lung damage, with potentially irreversible results. Little is known about the clinical aspects of this condition. Understanding its behavior could contribute to changing its potential devastating impact.

The objective of this study is to evaluate the incidence of VILI vortex in patients with acute respiratory syndrome (ARDS) secondary to COVID-19, to establish a connection between this phenomenon and mortality, and to identify the factors that have an impact on its development.

DETAILED DESCRIPTION:
Mechanical ventilation is an essential tool for the treatment of patients with acute respiratory distress syndrome (ARDS). However, as with other strategies, it is not free of complications. Inadequate ventilation may have a negative impact on pulmonary and systemic hemodynamics, and it could both cause structural damage to pulmonary parenchyma and activate inflammation (2). This process is known as ventilator-induced lung injury (VILI) and may promote the development of multiple organ failure and, eventually, death.

VILI results from the interaction between the mechanical load applied to the ventilable lung and its capacity to tolerate it. Factors such as tidal volume (Vt), driving pressure (ΔP), inspiratory flow rate (VI), respiratory rate (RR), excessive inspiratory effort, high levels of FiO2 and, in some cases, PEEP, have been involved in damage mechanism. In that sense, the concept of mechanical power (MP) tries to encompass most of these factors within a measurable unit (3). Furthermore, the decrease in ventilable lung volume (baby lung concept), the heterogeneous lung compromise in ARDS), and the presence of cofactors that have a negative impact on the lung (fluid overload, presence of sepsis or shock) could increase its susceptibility to damage (4-5).

Due to the fact that the mechanical conditions of the lung change dynamically with the progression of the disease, the ventilatory strategy needs constant adjustments in order to maintain a balance between the load and the size of the ventilable lung (concept of ergonomic ventilation). In fact, a protective ventilatory strategy of low tidal volume (Vt: 6 ml/kg/PBW) and limited plateau pressure (PPlat <30 cmH2O) may cause damage if the functional residual capacity (FRC) decreases significantly, thus making a lower number of alveoli (including capillaries) withstand a higher mechanical load per unit.

The concept of VILI vortex has recently been proposed as a progressive lung injury mechanism in which the alveolar stress/strain increases as the ventilable lung "shrinks". This positive feedback inexorably leads to the acceleration of lung damage, with potentially irreversible results (1). Little is known about the clinical aspects of this condition. Understanding its behavior could contribute to changing its potential devastating impact.

The objective of this study is to evaluate the incidence of VILI vortex in patients with ARDS secondary to COVID-19, to establish a connection between this phenomenon and mortality, and to identify the factors that have an impact on its development.

ELIGIBILITY:
Inclusion Criteria: ARDS

-

Exclusion Criteria:

Patients with do-not-resuscitate (DNR) orders and pregnant women. Cardiac arrest before ICU admission. Extra corporeal membrane oxygenation (ECMO) requirement within the first 24 h of ICU admission and chronic obstructive pulmonary disease with gold class 3 or 4, or home oxygen therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SARS-CoV-2 in mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Pistillo, Principal Investigator — Hospital El Cruce
Locations (1):
- Nestor Pistillo, Avellaneda, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marini JJ, Gattinoni L. Time Course of Evolving Ventilator-Induced Lung Injury: The "Shrinking Baby Lung". Crit Care Med. 2020 Aug;48(8):1203-1209. doi: 10.1097/CCM.0000000000004416. PMID 32697492
- [Background] Beitler JR, Malhotra A, Thompson BT. Ventilator-induced Lung Injury. Clin Chest Med. 2016 Dec;37(4):633-646. doi: 10.1016/j.ccm.2016.07.004. Epub 2016 Oct 14. PMID 27842744
- [Background] Gattinoni L, Pesenti A. The concept of "baby lung". Intensive Care Med. 2005 Jun;31(6):776-84. doi: 10.1007/s00134-005-2627-z. Epub 2005 Apr 6. PMID 15812622
- [Background] Gattinoni L, Tonetti T, Quintel M. Regional physiology of ARDS. Crit Care. 2017 Dec 28;21(Suppl 3):312. doi: 10.1186/s13054-017-1905-9. PMID 29297365
- [Background] Vasques F, Duscio E, Cipulli F, Romitti F, Quintel M, Gattinoni L. Determinants and Prevention of Ventilator-Induced Lung Injury. Crit Care Clin. 2018 Jul;34(3):343-356. doi: 10.1016/j.ccc.2018.03.004. PMID 29907269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between March 2020 to March 2021
Pre-assignment Details: No patients with SARS-CoV-2 were excluded from the study prior to group assignment.
Groups:
- VILI VORTEX: Clinical categorization of patients with SARS-CoV-2 with VILI vortex
- NO VILI VORTEX: Clinical categorization of patients with SARS-CoV-2 without VILI vortex
Period: Overall Study
Arm/Group | VILI VORTEX | NO VILI VORTEX
Started | 15 | 50
Completed | 15 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VILI VORTEX: Participants who evolved with VILI vortex clinical criteria
- No VILI VORTEX: Participants who evolved without clinical criteria for VILI vortex
- Total: Total of all reporting groups
Arm/Group | VILI VORTEX | No VILI VORTEX | Total
Number analyzed (Participants) | 15 | 50 | 65
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [55 to 60] | 60 [54 to 66] | 60 [55 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Percentage of male and female patients: Female | 6 | 18 | 24
  Percentage of male and female patients: Male | 9 | 32 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 50 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 15 | 50 | 65
Comorbidities [Number; unit: participants] — Risk factors at the time of admission
  participants
    Hypertension | 9 | 25 | 34
    Diabetes Mellitus | 25 | 33 | 58
    Obesity | 5 | 11 | 16
    Ischemic heart disease | 2 | 6 | 8
    COPD | 3 | 7 | 10
    Cancer/immunosupresion | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survived and Died
Description: The number of patients who died and survived was compared between patients with SARS-CoV-2 who progressed with VILI VORTEX and without VILI VORTEX)
Time Frame: 90 days
Population: The evolution of the patients was compared with Chi square, significant p <0.05
Measure: Count of Participants; unit: Participants
Groups:
- VILI VORTEX: Patients who evolved with clinical criteria of VILI VORTEX
- No VILI VORTEX: Patients who evolved without clinical criteria of VILI VORTEX
Arm/Group | VILI VORTEX | No VILI VORTEX
Number analyzed (Participants) | 15 | 50
Participants
  Survivors | 1 | 31
  Dead | 14 | 19

2. Primary Outcome: Number of Patients With and Without Refractory Hypoxemia
Description: The number of patients that evolved with refractory hypoxemia was compared between the patients with SARS-CoV-2 that evolved with VILI VORTEX and without VILI VORTEX) Refractory hypoxemia was defined as PaO2/FiO2 <100 despite the optimization of mechanical ventilation and prone positioning.
Time Frame: 90 days
Population: The baseline characteristics of the population were similar for both groups.
Measure: Number; unit: participants
Arm/Group | No VILI VORTEX | VILI VORTEX
Number analyzed (Participants) | 50 | 15
participants
  with refractory hypoxemia | 1 | 14
  no refractory hypoxemia | 49 | 1

3. Primary Outcome: Number of Patients With Complications
Description: The following variables and complications were also observed during the period of analysis: incidence of pneumonia associated with mechanical ventilation, need for noradrenaline over 0.1 γ/kg/min for more than 24 h, positive blood cultures, accumulated fluid balance, dialysis treatment, clinical and/or echocardiographic evidence of heart failure, lactate ≥2 mmol/L in at least two consecutive samples, presence of persistent fever (≥38º at least once a day for three consecutive days), and the highest value of ferritin, D-dimer, C-reactive protein, troponin I and LDH obtained during the first 14 days of invasive mechanical ventilation.
  VILI vortex patients had positive blood cultures, moderate to severe shock, persistent fever and fluid balance was considerably more positive.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | VILI VORTEX | No VILI VORTEX
Number analyzed (Participants) | 15 | 50
Participants
  intranosocomial pneumonia | 7 | 19
  Renal replacement therapy | 7 | 18
  Persistent fever | 7 | 10
  Bood cultures | 9 | 10

ADVERSE EVENTS:
Time Frame: up to 12 weeks after entering the study
Description: Refractory hypoxemia was defined as PaO2/FiO2 <100 despite the optimization of mechanical ventilation and prone positioning.
Groups:
- VILI VORTEX: SARS-CoV-2 patients who evolved with VILI VORTEX
- NO VILI VORTEX: SARS-CoV-2 patients who evolved without VILI VORTEX
Arm/Group | VILI VORTEX | NO VILI VORTEX
All-Cause Mortality (participants affected / at risk) | 14/15 | 19/50
Serious Adverse Events (participants affected / at risk) | 14/15 | 23/50
Other Adverse Events (participants affected / at risk) | 10/15 | 20/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VILI VORTEX (N=15) | NO VILI VORTEX (N=50)
Refractory hipoxemy (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 1 (1) — Refractory hypoxemia was defined as PaO2/FiO2 <100 despite the optimization of mechanical ventilation and prone positioning.
Severe Kidney Failure (Renal and urinary disorders) | 7 (7) | 18 (18) — AKI III: Increase in serum creatinine >300% from baseline or serum creatinine ≥4.0 mg/dl(≥354 umol/L) after an increase of at least 44 umol/L or treatment with renal replacement therapy.
Intranosocomial pneumonia (Infections and infestations) | 7 (7) | 19 (19)
Blood cultures (Infections and infestations) | 9 (9) | 10 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VILI VORTEX (N=15) | NO VILI VORTEX (N=50)
Lactate level >2mmol/L (Vascular disorders) | 7 (7) | 16 (16) — Lactate level> 2 mmol / L is associated with shock
Persistent fever (General disorders) | 7 (7) | 10 (10) — Tº >37.9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT04174313/Prot_SAP_000.pdf